CLINICAL TRIAL: NCT04092751
Title: An Open-Label, Randomized, Two- Period Crossover Study to Evaluate the Effect of Oral Doses of SCY-078 (Ibrexafungerp) on the Pharmacokinetics of Pravastatin Administered Orally to Healthy Subjects
Brief Title: Study to Evaluate the Effect of SCY-078 (Ibrexafungerp) on the PK of Pravastatin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Collaborators: Clinical Network Services (CNS) Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SCY-078-115
Record Dates: First submitted 2019-09-10; First posted 2019-09-17 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Pharmacokinetics
Keywords: SCY-078; Ibrexafungerp; Pravastatin; Healthy Subjects; Pharmacokinetics
MeSH Terms: interventions — ibrexafungerp

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to a treatment sequence (AB or BA) in a crossover fashion with a minimum 10-day washout period between treatments
  Treatment A = Single oral 20-mg dose of PRA on Day 1 AM. Treatment B = Twice daily (BID), every 12 hours (Q12H) oral doses of SCY-078 750 mg on Day 1 and Day 2; and on Day 3 a single AM dose of oral SCY 078 750 mg followed by a single 20-mg dose of PRA administered one hour later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Single oral 20-mg dose of PRA on Day 1 AM
  Interventions: Drug: PRA
- Treatment B (Experimental): Twice daily (BID), every 12 hours (Q12H) oral doses of SCY-078 750 mg on Day 1 and Day 2; and on Day 3 a single AM dose of oral SCY 078 750 mg followed by a single 20-mg dose of PRA administered one hour later.
  Interventions: Drug: SCY-078 plus PRA

INTERVENTIONS:
Drug: PRA — Single oral 20-mg dose of PRA on Day 1 AM
  Arms: Treatment A
Drug: SCY-078 plus PRA — Twice daily (BID), every 12 hours (Q12H) oral doses of SCY-078 750 mg on Day 1 and Day 2; and on Day 3 a single AM dose of oral SCY 078 750 mg followed by a single 20-mg dose of PRA administered one hour later
  Arms: Treatment B

SUMMARY:
This is an Open-Label, Randomized, Two-Period, Crossover Study to Evaluate the Effect of Oral Doses of SCY-078 (Ibrexafungerp) on the Pharmacokinetics of Pravastatin Administered Orally to Healthy Subjects

DETAILED DESCRIPTION:
The two period crossover study will consist of two treatments administered in random order separated by a minimum 10 day washout interval (between the last dose in the first period and the first dose in the subsequent period).

28 healthy adult male and female subjects will be enrolled to determine the effects of SCY-078 on the pharmacokinetics of a single-dose of PRA.

Subjects will undergo a screening visit 4 weeks prior to dosing.

Subjects will be randomized to a treatment sequence (AB or BA) in a crossover fashion:

Treatment A = Single oral 20-mg dose of PRA on Day 1 AM.

Treatment B = Twice daily (BID) oral doses of SCY-078 750 mg (5 X 150-mg tablets) on Day 1 and Day 2; and on Day 3 a single AM dose of oral SCY 078 750 mg followed one hour later by a single 20-mg oral dose of PRA.

All subjects will be admitted to the clinical site on Day -1 in each period and will then fast overnight and will stay in the clinical site until the final procedures are performed in that treatment period, and then they may be discharged.

For Treatment B, on Day 1, 2, and 3, limited PK blood samples will be collected for SCY 078 assays.

For Treatments A on Days 1 and 2, and Treatment B on Day 3, serial PK blood samples will be collected for PRA assays.

ELIGIBILITY:
Inclusion Criteria:

1. is a male or female between 18 to 55 years, inclusive, of age at the prestudy (screening) visit (time of signing the Informed Consent).
2. has a Body Mass Index (BMI) 18.0 to 32 kg/m2 at the prestudy (screening) visit.
3. is judged to be in good health based on medical history, physical examination, vital sign measurements, electrocardiogram (ECG), and laboratory safety tests performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug.
4. has been is a nonsmoker and/or has not used nicotine or nicotine-containing products for approximately 6 months prior to screening.
5. is willing and able to understand and provide signed informed consent and understands the study procedures and agrees to participate in the study.
6. is not pregnant or lactating (for women of childbearing potential) and must agree to use adequate double barrier birth control.

NOTE: Women of childbearing potential must have a negative serum pregnancy test (β human chorionic gonadotropin [β-hCG]) at Screening visit and negative urine pregnancy test at each treatment period (conducted on Day -1 prior to dosing).

Exclusion Criteria:

1. has a contra-indication to Pravachol® (pravastatin sodium).
2. has severe liver disease or chronically elevated liver enzymes.
3. is pregnant or lactating
4. has a history of uncontrolled or unstable cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematopoietic, neoplastic, and/or neurological disease.
5. has a current or recent (within 3 months) gastrointestinal (GI) disease or any GI surgery that could impact absorption of study drug.
6. has a history of any illness that, in the opinion of the investigator, could confound the results of the study or pose an additional risk to the subject by their participation in the study.
7. has a QTcF interval >480 msec at the Screening or Day -1 visits of the study.
8. subject consumed Seville or blood oranges, grapefruit or grapefruit juice, or mulberry juice , as well as vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard) and or charbroiled meats from 4 days prior to the dose of study medication.
9. has consumed any alcohol within 7 days before dosing SCY-078 prior to dose of study medication or has a history of alcohol abuse.
10. has a positive drug and or alcohol screen at screening and or (each) admission to the clinical research center.
11. is a smoker or has used tobacco or any nicotine-containing products within the 6 months prior to the first dosing in the study screening.
12. has been participated in a clinical investigation of any drug, biological, or other investigational therapy, device or procedure 30 days before dosing
13. has a history of an allergic reaction to SCY-078 or any of its excipients, or is allergic to Pravachol® (pravastatin sodium), or its inactive ingredients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of PRA administered with SCY-078, AUC | 24 days
  AUC 0-24 of PRA when taken with SCY-078.

SECONDARY OUTCOMES:
Pharmacokinetics of PRA administered with SCY-078, Cmax | 24 days
  Cmax PRA when taken with SCY-078
Pharmacokinetics of PRA administered with SCY-078, Tmax | 24 days
  Tmax of PRA when taken with SCY-078.
Pharmacokinetics of PRA administered with SCY-078, Half life (t1/2) | 24 days
  Half life (t1/2) of PRA when taken with SCY-078.
Safety and tolerability of oral dosing of combination of PRA with SCY-078 | 6 weeks
  Incidence of treatment-related adverse events (AE) and discontinuations due to (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Scientia Clinical Research Limited Bright Building, Randwick, New South Wales, Australia